CLINICAL TRIAL: NCT04561219
Title: Nitazoxanide for Moderate to Severe COVID-19 Pneumonia: a Multicenter, Randomized, Placebo-controlled, Double-Blind Clinical Trial
Brief Title: Nitazoxanide Therapy for Patients With COVID-19 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Ministry of Science and Technology, Brazil (Other); National Research Council, Brazil (Other); Financiadora de Estudos e Projetos (Other); ATCGen (Unknown); Hospital Central da Aeronáutica, Rio de Janeiro (Unknown); Hospital da Força Aérea do Galeão (Unknown); Hospital Naval Marcilio Dias (Unknown); Hospital Universitario Pedro Ernesto (Other); Hospital de Força Aérea de São Paulo (Unknown); Hospital das Clínicas Luzia de Pinho Melo (Unknown); Complexo Hospitalar Municipal de São Caetano do Sul (Unknown); Hospital Municipal de Barueri Dr Francisco Moran (Unknown); Hospital Regional de Sorocaba Dr Adib Domingos Jatene (Unknown); Hospital Geral de São Mateus Dr Manoel Bifulco (Unknown); Santa Casa de Misericórdia de Belo Horizonte (Other); Mater Dei Hospital, Brazil (Other); Hospital Eduardo de Menezes (Unknown); Hospital das Clínicas da Universidade Federal de Pernambuco (Unknown); Hospital das Forças Armadas, Brazil (Other); Hospital Regional da Asa Norte, Brazil (Unknown); Complexo Hospitalar do Trabalhador de Curitiba (Unknown); Hospital Estadual de Doenças Tropicais Dr Anuar Auad (Unknown); Hospital Geral de Fortaleza (Other Government)
Responsible Party: Principal Investigator, Jose Roberto Lapa e Silva, Clinical Investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SARITA-1; RBR-88bs9x (Other: Registro Brasileiro de Ensaios Clínicos (REBEC)); 30662420.0.1001.0008 (Other: Comitê Nacional de Ética em Pesquisa (CONEP))
Record Dates: First submitted 2020-09-22; First posted 2020-09-23 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Corona Virus Infection; Pneumonia, Viral
Keywords: covid19; coronavirus; clinical trial; placebo-controlled; randomized; brazil; nitazoxanide; hospitalized patients; covid-19; sars-cov-2; new coronavirus; multicenter; double-blind
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Pneumonia, Viral | interventions — nitazoxanide

STUDY DESIGN:
Intervention Model Description: Hospitalized patients with clinical signs of COVID-19, and either chest tomography scans suggestive of COVID-19 or confirmed by RT-PCR molecular tests, will be randomly divided into 2 groups: experimental and control groups.
  Experimental group: 250 hospitalized patients diagnosed with COVID-19 derived pneumonia will receive nitazoxanide 500mg 8/8 hs for 5 days. Control group: 250 hospitalized patients diagnosed with COVID-19 derived pneumonia will receive placebo 8/8 hs for 5 days.
Who Masked: Participant, Care Provider
Masking Description: Patients were randomly allocated into one of the two groups: A or B. Patients received labelled medication: A or B, by the pharmacist. Patients received an identification number, so care providers, outcomes assessors and investigators did not know anything regarding the patients' groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Experimental): Patients received nitazoxanide 500mg 8/8hours, for 5 days.
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): Patients received placebo 500mg 8/8hours, for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide 500mg three times a day for 5 days
  Other Names: annita; azox; irose; tanisea; trinida; zoxany
  Arms: Nitazoxanide
Drug: Placebo — Placebo three times a day for 5 days
  Arms: Placebo

SUMMARY:
Multicenter, randomized, placebo-controlled, parallel, blinded, interventional, treatment clinical trial with two arms.

Population: 500 Hospitalized patients with pneumonia derived from COVID-19 (Coronavirus Disease-19), either confirmed by RT-PCR (Real Time polymerase chain reaction), or suggested by typical findings on the computed tomography scan symptomatic.

Experimental group: nitazoxanide 500mg 8 / 8 hours for 5 days. Control group: placebo 8/8 hours for 5 days.

DETAILED DESCRIPTION:
SARITA-1 is a multicenter, randomized, placebo-controlled, parallel, blinded, interventional, treatment clinical trial with two arms, which aims to study the impact of nitazoxanide for hospitalized patients with pneumonia derived from COVID-19 (Coronavirus Disease-19) Experimental group: 250 patients received nitazoxanide 500mg 8 / 8 hours for 5 days. Control group: 250 patients received placebo 8/8 hours for 5 days.

Population: Patients with clinical symptoms of COVID-19: dyspnoea and/or fever and/or cough) and: either computed tomography scan suggestive of viral pneumonia or confirmatory molecular test by RT-PCR (Real Time polymerase chain reaction),

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring supplemental oxygen [peripheral oxygen saturation (SpO2) < 93%], admitted to hospital with COVID-19 symptoms associated with chest computed tomography (CT) scan suggestive of viral pneumonia or positive nasopharyngeal swab test for SARS-CoV2 (RT-PCR)
* Age equal or superior to 18 years
* Non-pregnant women
* Willingness to receive study treatment
* Providing written and informed consent or the same consent signed by a family member

Exclusion Criteria:

* Impossibility to use oral medications
* History of severe liver disease (Child Pugh C class)
* Previous renal failure
* Severe heart failure (NYHA 3 or 4)
* COPD (GOLD 3 and 4)
* Neoplasia in the last 5 years
* Known autoimmune disease
* Individuals with known hypersensitivity to study drug
* Previous treatment with the study medication during the last 30 days
* Clinical suspicion of tuberculosis and bacterial pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-04-19 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Orotracheal intubation rate | 14 days
  Compare the intubation rate of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, in the period of 14 days; verified by clinical evolution; quantified by percentage.

SECONDARY OUTCOMES:
Hospitalisation days | 14 days
  Compare the number of days patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, stayed at the hospital, in the period of 14 days; verified by clinical evolution; quantified by absolute number.
ICU days | 14 days
  Compare the number of days patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, stayed at the ICU, in the period of 14 days; verified by clinical evolution; quantified by absolute number.
Intranasal oxygen support days | 14 days
  Compare the number of days patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, stayed with the support of oxygen nasal cannula, in the period of 14 days; verified by clinical evolution; quantified by absolute number.
Mortality rate | 14 days
  Compare the mortality rate of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, in the period of 14 days; verified by clinical evolution; quantified by absolute number.
Days with fever | 14 days
  Reduction in the duration of fever of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide compared to patients treated with placebo; verified through the collection of clinica data; quantified by the number of days that presented the symptom.
Days with cough | 14 days
  Reduction in the duration of cough of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide compared to patients treated with placebo; verified through the collection of clinica data; quantified by the number of days that presented the symptom.
Days with dyspnea | 14 days
  Reduction in the duration of dyspnea of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide compared to patients treated with placebo; verified through the collection of clinica data; quantified by the number of days that presented the symptom.
Radiologic findings | Day1
  Compare chest tomographic findings of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide compared to patients treated with placebo; verified through the collection of radiologic data; quantified by the number of patients that presented the a list of alterations.
Radiologic findings | Day7
  Compare chest tomographic findings of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide compared to patients treated with placebo; verified through the collection of radiologic data; quantified by the number of patients that presented the a list of alterations.
Cardiologic findings | Day1
  Compare echocardiographic findings of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide compared to patients treated with placebo; verified through the collection of echocardiographic data; quantified by the number of patients that presented the a list of alterations.
Cardiologic findings | Day7
  Compare echocardiographic findings of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide compared to patients treated with placebo; verified through the collection of echocardiographic data; quantified by the number of patients that presented the a list of alterations.
C-reactive protein - absolute number | Day 1
  To evaluate the levels of C-reactive protein (CRP) of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 1; verified by laboratory tests and expressed by the absolute number between the two groups.
C-reactive protein serum levels | Day 3
  To evaluate the levels of C-reactive protein (CRP) of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
C-reactive protein serum levels | Day 7
  To evaluate the levels of C-reactive protein (CRP) of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 7; verified by laboratory tests and expressed by the absolute number between the two groups.
Lactate dehydrogenase (LDH) serum levels | Day 1
  To evaluate the levels of lactate dehydrogenase (LDH) of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 1; verified by laboratory tests and expressed by the absolute number between the two groups.
Lactate dehydrogenase (LDH) serum levels | Day 3
  To evaluate the levels of lactate dehydrogenase (LDH) of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
Lactate dehydrogenase (LDH) serum levels | Day 7
  To evaluate the levels of lactate dehydrogenase (LDH) of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 7; verified by laboratory tests and expressed by the absolute number between the two groups.
Troponin serum levels | Day 1
  To evaluate the levels of troponin of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 1; verified by laboratory tests and expressed by the absolute number between the two groups.
Troponin serum levels | Day 3
  To evaluate the levels of troponin of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
Troponin serum levels | Day 7
  To evaluate the levels of troponin of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 7; verified by laboratory tests and expressed by the absolute number between the two groups.
Electrolytes serum levels | Day 1
  To evaluate the levels of electrolytes of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 1; verified by laboratory tests and expressed by the absolute number between the two groups.
Electrolytes serum levels | Day 3
  To evaluate the levels of electrolytes of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
Electrolytes serum levels | Day 7
  To evaluate the levels of electrolytes of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 7; verified by laboratory tests and expressed by the absolute number between the two groups.
Glucose serum levels | Day 1
  To evaluate the levels of glucose of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 1; verified by laboratory tests and expressed by the absolute number between the two groups.
Glucose serum levels | Day 3
  To evaluate the levels of glucose of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
Glucose serum levels | Day 7
  To evaluate the levels of glucose of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 7; verified by laboratory tests and expressed by the absolute number between the two groups.
Renal function | Day 1
  To evaluate renal function of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 1; verified by laboratory tests and expressed by the absolute number between the two groups.
Renal function | Day 3
  To evaluate renal function of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
Renal function | Day 7
  To evaluate renal function of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 7; verified by laboratory tests and expressed by the absolute number between the two groups.
Coagulogram | Day 1
  To evaluate coagulogram of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 1; verified by laboratory tests and expressed by the absolute number between the two groups.
Coagulogram | Day 3
  To evaluate coagulogram of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
Coagulogram | Day 7
  To evaluate coagulogram of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 7; verified by laboratory tests and expressed by the absolute number between the two groups.
Liver function panel | Day 1
  To evaluate liver function panel of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 1; verified by laboratory tests and expressed by the absolute number between the two groups.
Liver function panel | Day 3
  To evaluate liver function panel of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
Liver function panel | Day 7
  To evaluate liver function panel of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 7; verified by laboratory tests and expressed by the absolute number between the two groups.
Ferritin | Day 1
  To evaluate ferritin of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 1; verified by laboratory tests and expressed by the absolute number between the two groups.
Ferritin | Day 3
  To evaluate ferritin of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
Ferritin | Day 7
  To evaluate ferritin of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 7; verified by laboratory tests and expressed by the absolute number between the two groups.
D-dimer | Day 1
  To evaluate D-dimer of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 1; verified by laboratory tests and expressed by the absolute number between the two groups.
D-dimer | Day 3
  To evaluate D-dimer of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
D-dimer | Day 7
  To evaluate D-dimer of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 7; verified by laboratory tests and expressed by the absolute number between the two groups.
Blood cell count | 7 days
  To evaluate blood cell count of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, for 7 days; verified by laboratory tests and expressed by the absolute number between the two groups.
Inflammatory mediators | Day 1
  To evaluate D-dimer of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 1; verified by laboratory tests and expressed by the absolute number between the two groups.
Inflammatory mediators | Day 3
  To evaluate D-dimer of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 3; verified by laboratory tests and expressed by the absolute number between the two groups.
Inflammatory mediators | Day 7
  To evaluate D-dimer of patients with COVID-19 submitted to the therapeutic protocol with nitazoxanide with patients with COVID-19 treated with placebo, on day 7; verified by laboratory tests and expressed by the absolute number between the two groups.

OTHER OUTCOMES:
Adverse events - percentage | Day 14
  Assess the incidence and profile of adverse events reported throughout the study, by treatment group; verified by information actively collected from patients or family members; quantified by percentage.
Adverse events - absolute number | Day 14
  Assess the incidence and profile of adverse events reported throughout the study, by treatment group; verified by information actively collected from patients or family members; quantified by absolute number.
Treatment discontinuation rate - absolute number | Day 14
  Assess the rate of treatment discontinuation due to adverse events; verified by information actively collected from patients or family members; quantified by absolute number.
Treatment discontinuation rate - percentage | Day 14
  Assess the rate of treatment discontinuation due to adverse events; verified by information actively collected from patients or family members; quantified by percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro L Silva, PhD, Study Chair — Universidade Federal do Rio de Janeiro; Patricia RM Rocco, MD, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan on sharing all IPD that underlie results in a publication for editorial board, with cautious of not sharing confidential data.
Supporting Information: Study Protocol, SAP
Time Frame: Available as soon as the editorial board of the journal accepting the manuscript requires.
Access Criteria: Editorial board of the Journal accepting the manuscript.

REFERENCES:
- [Background] Rossignol JF. Nitazoxanide, a new drug candidate for the treatment of Middle East respiratory syndrome coronavirus. J Infect Public Health. 2016 May-Jun;9(3):227-30. doi: 10.1016/j.jiph.2016.04.001. Epub 2016 Apr 16. PMID 27095301
- [Background] Rossignol JF. Nitazoxanide: a first-in-class broad-spectrum antiviral agent. Antiviral Res. 2014 Oct;110:94-103. doi: 10.1016/j.antiviral.2014.07.014. Epub 2014 Aug 7. PMID 25108173
- [Background] Rajoli RK, Pertinez H, Arshad U, Box H, Tatham L, Curley P, Neary M, Sharp J, Liptrott NJ, Valentijn A, David C, Rannard SP, Aljayyoussi G, Pennington SH, Hill A, Boffito M, Ward SA, Khoo SH, Bray PG, O'Neill PM, Hong WD, Biagini G, Owen A. Dose prediction for repurposing nitazoxanide in SARS-CoV-2 treatment or chemoprophylaxis. medRxiv [Preprint]. 2020 May 6:2020.05.01.20087130. doi: 10.1101/2020.05.01.20087130. PMID 32511548
- [Background] Pepperrell T, Pilkington V, Owen A, Wang J, Hill AM. Review of safety and minimum pricing of nitazoxanide for potential treatment of COVID-19. J Virus Erad. 2020 Apr 30;6(2):52-60. doi: 10.1016/S2055-6640(20)30017-0. PMID 32405422
- [Derived] Conceicao CCS, Martins CM, Medeiros Silva M, Neto HCCF, Chiumello D, Rocco PRM, Cruz FF, Silva PL. Predicting clinical outcomes at hospital admission of patients with COVID-19 pneumonia using artificial intelligence: a secondary analysis of a randomized clinical trial. Front Med (Lausanne). 2025 May 2;12:1561980. doi: 10.3389/fmed.2025.1561980. eCollection 2025. PMID 40385586
- [Derived] Silva PL, Cruz FF, Martins CM, Herrmann J, Gerard SE, Xin Y, Cereda M, Ball L, Pelosi P, Rocco PRM. A specific combination of laboratory data is associated with overweight lungs in patients with COVID-19 pneumonia at hospital admission: secondary cross-sectional analysis of a randomized clinical trial. Front Med (Lausanne). 2023 May 16;10:1137784. doi: 10.3389/fmed.2023.1137784. eCollection 2023. PMID 37261117
- [Derived] Rocco PRM, Silva PL, Cruz FF, Tierno PFGMM, Rabello E, Junior JC, Haag F, de Avila RE, da Silva JDG, Mamede MMS, Buchele KS, Barbosa LCV, Cabral AC, Junqueira AAF, Araujo-Filho JA, da Costa LATJ, Alvarenga PPM, Moura AS, Carajeleascow R, de Oliveira MC, Silva RGF, Soares CRP, Fernandes APSM, Fonseca FG, Camargos VN, Reis JS, Franchini KG, Luiz RR, Morais S, Sverdloff C, Martins CM, Felix NS, Mattos-Silva P, Nogueira CMB, Caldeira DAF, Pelosi P, Lapa-E-Silva JR. Nitazoxanide in Patients Hospitalized With COVID-19 Pneumonia: A Multicentre, Randomized, Double-Blind, Placebo-Controlled Trial. Front Med (Lausanne). 2022 Apr 13;9:844728. doi: 10.3389/fmed.2022.844728. eCollection 2022. PMID 35492335